CLINICAL TRIAL: NCT03447054
Title: Treating Alcohol Dependence : Testing a Combined Treatment Model Using Transcranial Direct Current Stimulation (tDCS) and Inhibitory Control Training (ICT)
Brief Title: Severe Alcohol-use Disorder: a tDCS and Response Inhibition Training Intervention
Acronym: ALCOSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Collaborators: University Ghent (Other); Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Xavier NOËL, Research Associate at the F.R.S/FNRS, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Baudoin_2016_J1130650_206500
Record Dates: First submitted 2017-11-03; First posted 2018-02-27 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; tDCS; inhibition; cognitive training; implicit cognition; relapse; craving
MeSH Terms: conditions — Alcoholism; Inhibition, Psychological; Recurrence | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 2 (active, sham tDCS) x 2 (active, inactive response inhibition training) factorial design
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combined TDCS active and ICT active (Experimental): Five consecutive days: Twenty minutes of TDCS on the right dorsolateral prefrontal cortex while performing an alcohol-cue inhibitory control training consisting to systematically paired go responses with non-alcohol pictures and no-go responses with alcohol-related pictures.
  Interventions: Behavioral: Combined TDCS active and ICT active
- Combined TDCS sham and ICT active (Active Comparator): Five consecutive days: Twenty minutes of sham TDCS on the right dorsolateral prefrontal cortex, while performing a no-cue go/no-go training consisting to carry out a go/no-go paradigm with no alcohol-related content.
  Interventions: Behavioral: Combined Sham TDCS and inactive ICT
- Combined TDCS active and ICT inactive (Active Comparator): Five consecutive days: Twenty minutes of active TDCS in association with no-cue go/no-go training consisting to carry out a go/no-go paradigm with no alcohol-related content.
  Interventions: Behavioral: Combined TDCS active and ICT inactive
- Combined Sham TDCS and inactive ICT (Sham Comparator): Five consecutive days: Twenty minutes of Inactive TDCS combined with an non alcohol-cue inhibitory control training consisting to carry out a go/no-go paradigm with no alcohol-related content.
  Interventions: Behavioral: Combined TDCS sham and ICT active

INTERVENTIONS:
Behavioral: Combined TDCS active and ICT active — Five 20-minute long sessions including TDCS (2 MicroAmperes during 20 minutes) and ICT, 5 consecutive days
  Other Names: Experimental
  Arms: Combined TDCS active and ICT active
Behavioral: Combined TDCS sham and ICT active — Five 20-minute long sessions including TDCS sham (non active) and ICT, 5 consecutive days
  Other Names: Sham/active
  Arms: Combined Sham TDCS and inactive ICT
Behavioral: Combined TDCS active and ICT inactive — Five 20-minute long sessions including TDCS sham and no-cue inhibition training, 5 consecutive days
  Other Names: Sham/inactive
  Arms: Combined TDCS active and ICT inactive
Behavioral: Combined Sham TDCS and inactive ICT — Five 20-minute long sessions including TDCS and no-cue inhibition training, 5 consecutive days
  Other Names: Active/inactive
  Arms: Combined TDCS sham and ICT active

SUMMARY:
Most severe forms of alcohol-use disorder are thought to reflect an abnormal interplay between two neural systems: an overly active impulsive one driven by immediate rewards prospects and a weak reflective one, tuned on long-term prospects. The investigators propose that two non-pharmacological interventions, Transcranial Direct Current Stimulation (tDCS) and Inhibitory Control Techniques (ICT) may act on both systems when combined, which might ultimately result is a reduction of alcohol relapse rate.

DETAILED DESCRIPTION:
Treating Alcohol dependence remains notoriously difficult despite use of several medications, psychotherapeutic and psychosocial interventions. Alcohol dependence is thought to reflect an abnormal interplay between two neural systems: an overly active impulsive one driven by immediate rewards prospects and a weak reflective one, tuned on long-term prospects. The investigators proposes that two non-pharmacological interventions, Transcranial Direct Current Stimulation (tDCS) and Inhibitory Control Techniques (ICT) may act on both systems when combined. tDCS has been found to improve working memory, which is necessary to evaluate long-term consequences of actions. ICT is able to modify the automatic approach tendencies towards appetitive cues.

The investigators will recruit 160 alcohol-dependent patients and divide them randomly between four treatment conditions : real transcranial Direct Current Stimulation (tDCS) with active or control Inhibitory Control Technique (ICT ); or sham (placebo) tDCS with active or control ICT.

Patients will be evaluated with primary outcome measures (alcohol consumption patterns) and secondary outcome measures (working memory and changes in alcohol-related stimuli affective values).

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe alcohol-use disorder (DSM-5 criteria), hospitalized for detoxification.
* Severity of alcohol use disorder must be at least moderate (at least 4 DSM-5 criteria)
* Aged between 18 and 65 years
* Comorbidity with anxiety disorders and depressive disorders is allowed
* Patients must be illegal drug free for 3 weeks at beginning of trial
* Pharmacotherapy: patients should be benzodiazepines free at the moment of inclusion. They are allowed to continue other psychotropic medication (antidepressants, antipsychotics, mood stabilizers), providing they are following a stable regimen that will not be changed during the protocol time.
* Patients must be reachable for follow-up

Exclusion Criteria:

* Previous neurological conditions (epilepsy, traumatic brain injury, stroke)
* Present delirium, confusion or severe cognitive disorder
* Schizophrenia, chronic psychotic disorders, bipolar type 1 disorder.
* Any severe, life-threatening disorders
* High suicidal risk
* Specific contraindications for tDCS: metallic plates in the head
* Alcohol medication treatment initiated during the rehab: acamprosate, disulfiram, baclofen, nalmefen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Reduction of alcohol use in post-treatment at week 2 | é weeks post-rehab
  Based on self-report questionnaires (grams of ethanol/occasion, per/day, number of consecutive days of alcohol drinking)
Reduction of alcohol use in post-treatment at week 4 | 4 weeks post-rehab
  Based on self-report questionnaires (grams of ethanol/occasion, per/day, number of consecutive days of alcohol drinking)
Reduction of the relapse rate in post-treatment at week 2 | 2 weeks post-rehab
  Based on self-report questionnaires and on one other significant person's feedback; binary outcome (relapser or non-relapser)
Reduction of the relapse rate in post-treatment at week 4 | 4 weeks post-rehab
  Based on self-report questionnaires and on one other significant person's feedback; binary outcome (relapser or non-relapser)
Reduction of alcohol use in post-treatment at week 12 | 12 weeks post-rehab
  Based on self-report questionnaires (grams of ethanol/occasion, per/day, number of consecutive days of alcohol drinking)
Reduction of the relapse rate in post-treatment at week 12 | 12 weeks post-rehab
  Based on self-report questionnaires and on one other significant person's feedback; binary outcome (relapser or non-relapser)
Reduction of alcohol use in post-treatment at week 24 | 24 weeks post-rehab
  Based on self-report questionnaires (grams of ethanol/occasion, per/day, number of consecutive days of alcohol drinking)
Reduction of the relapse rate in post-treatment at week 24 | 24 weeks post-rehab
  Based on self-report questionnaires and on one other significant person's feedback; binary outcome (relapser or non-relapser)

SECONDARY OUTCOMES:
Cue reactivity (attractiveness) at day 22 | at post-intervention (day 22 of hospitalization)
  measures of attractiveness of used and novel alcohol-related pictures: Likert scale ranging from not (score of 0) at all to very much (score of 9)
Cue reactivity at day 22 | at post-intervention (day 22 of hospitalization)
  measures of attractiveness of used and novel alcohol-related pictures: Likert scale ranging from not (score of 0) at all to very much (score of 9)
Cue reactivity (valence) at day 22 | at post-intervention (day 22 of hospitalization)
  emotional content (valence) of pictures used in the response inhibition practice and of new pictures. Likert scale ranging from not (score of 0) at all to very much (score of 9)
Cue reactivity (arousal) at day 22 | at post-intervention (day 22 of hospitalization)
  emotional content (arousal) of pictures used in the response inhibition practice and of new pictures. Likert scale ranging from not (score of 0) at all to very much (score of 9)
Cue reactivity (alcohol verbal fluency) at day 12 | at baseline (day 12 of hospitalization)
  Alcohol verbal fluency (from Goldstein et al., 2007; Drug and Alcohol Dependence, 89:97-101 and Hon et al., 2016, Psychopharmacology, 233: 851-861: Participants are instructed to name as many alcohol-related words as possible in 1 min. Responses were audio recorded and independently coded into three categories: neutral, positive and negative valence by two researchers.
Cue reactivity (alcohol verbal fluency) at day 22 | at post-intervention (day 22 of hospitalization)
  Alcohol verbal fluency (from Goldstein et al., 2007; Drug and Alcohol Dependence, 89:97-101 and Hon et al., 2016, Psychopharmacology, 233: 851-861: Participants are instructed to name as many alcohol-related words as possible in 1 min. Responses were audio recorded and independently coded into three categories: neutral, positive and negative valence by two researchers.
response inhibition at day 12 | at baseline (day 10 of hospitalization)
  stop signal task (Logan, 1994): Stop Signal Reaction Time measure
response inhibition at day 22 | at post-intervention (day 22 of hospitalization)
  stop signal task (Logan, 1994): Stop Signal Reaction Time measure

CONTACTS AND LOCATIONS:
Locations (1):
- CHU-Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dubuson M, Kornreich C, Vanderhasselt MA, Baeken C, Wyckmans F, Dousset C, Hanak C, Veeser J, Campanella S, Chatard A, Jaafari N, Noel X. Transcranial direct current stimulation combined with alcohol cue inhibitory control training reduces the risk of early alcohol relapse: A randomized placebo-controlled clinical trial. Brain Stimul. 2021 Nov-Dec;14(6):1531-1543. doi: 10.1016/j.brs.2021.10.386. Epub 2021 Oct 20. PMID 34687964
- See also: PI researchgate profile — https://www.researchgate.net/profile/Xavier_Noel